CLINICAL TRIAL: NCT00842972
Title: Is Carotid Intima-media Thickness Affected by A1C Variability?
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Ahn, Chul Woo, Gangnam Severance Hospital
Other Study IDs: 3-2006-0005
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Type 2 Diabetes; A1C Variability
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study was conducted to evaluate the effect of A1C variability on the progression of carotid artery intima-media thickness in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* type II
* fluoroscopy in carotid once a year during 2 years

Exclusion Criteria:

* type 1 diabetes
* history or clinical evidence of coronary artery disease or cerebral or peripheral vascular disease
* the presence of albuminuria (defined as 24 hour urine albumin excretion ≥ 30 mg)
* renal dysfunction (defined as creatinine blood level ≥ 2.0 mg/dL)
* hepatic dysfunction (defined as alanine aminotransferase and/or aspartate aminotransferase blood level ≥ 3 × upper normal limit)
* smoking within the past 3 months prior to commencement of the study
* use of any medication likely to alter IMT such as calcium channel blocker, thiazolidinedione, antiplatelet agent (clopidogrel, cilostazol)
* use of glucocorticoid
* pregnancy
* severe concomitant disease such as cancer
* infection
* Cushing's syndrome
* acromegaly, or any other disorder likely to alter glycemia
* primary hypercholesterolemia
* hypothyroidism or hyperthyroidism
* use of any hormonal drugs
* alcoholism or drug abuse

Ages: 34 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: typeII, Fluroscopy in carotid once a year during 2 years.
Sampling Method: Probability Sample